CLINICAL TRIAL: NCT00372528
Title: An Open-Label, Multi-Center, Add-On Study Of Pregabalin (LYRICA) In Subjects With Refractory Partial Seizures Who Have Completed Studies 1008-010, 1008-035, 1008-114 Or 1008-164
Brief Title: An Open-Label Study Of Pregabalin In Subjects With Refractory Partial Seizures
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was terminated on April 8, 2011 as Pfizer Canada could no longer supply study drug. No efficacy or safety concerns factored into this decision.
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0081140
Record Dates: First submitted 2006-09-05; First posted 2006-09-07 (Estimated); Results first posted 2012-10-23 (Estimated); Last update posted 2021-01-26 (Actual); Status verified 2012-09

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pregabalin (Experimental): open label treatment
  Interventions: Drug: pregabalin (LYRICA)

INTERVENTIONS:
Drug: pregabalin (LYRICA) — 150 mg up to a maximum of 600 mg per day bid or tid as required

SUMMARY:
The main purpose of this trial is to allow continued access to pregabalin to Canadian subjects who participated in global pregabalin epilepsy studies 1008-010; 1008-035; 1008-114 and 1008-164 and to continue to study the long term safety of pregabalin administered as adjunctive therapy at dosages from 150 mg/day to 600 mg/day in Canadian subjects with refractory partial seizures.

ELIGIBILITY:
Inclusion Criteria:

* Must have completed Pfizer open-label studies 1008-010; 1008-035; 1008-114 or 1008-164 and wishes to continue receiving open-label pregabalin
* Must have responded favorably to pregabalin in Pfizer open-label study 1008-010, 1008-035, 1008-114 or 1008-164 and in the clinical opinion of the investigator continued treatment with pregabalin is in the the patient's best medical interest

Exclusion Criteria:

* Is pregnant or is considering becoming pregnant during the course of the study
* Experienced a serious adverse event during open-label Pfizer study 1008-010, 1008-035, 1008-114 or 1008-164

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- Canada (5):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, Barrie, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Windsor, Ontario

RESULTS

PARTICIPANT FLOW:
Groups:
- Pregabalin: Pregabalin 150 to 600 milligram (mg) capsule orally twice daily, as per investigator's discretion. Treatment was administered continuously as long as therapeutic response and tolerability was maintained, up to 5 years.
Period: Overall Study
Arm/Group | Pregabalin
Started | 21
Completed | 0
Not Completed | 21
Not completed — Lack of Efficacy | 1
Not completed — Adverse Event | 1
Not completed — Study Terminated by Sponsor | 18
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pregabalin
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.0 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 9
Mean Number of Seizures [Mean (Standard Deviation); unit: Seizures] — Seizures were episodes of disturbed brain activity that cause changes in attention or behavior. The different types of seizures observed were complex partial, secondarily generalized tonic-clonic, simple partial and others. Mean number of seizures were calculated from baseline visit to 1 day before Month 6 visit.
  Seizures | 30.70 (40.63)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 30 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to Year 5 and follow-up (30 days after last dose)
Population: Safety Analysis Set (SAS) included all participants who had received at least 1 dose of study medication in the open label period.
Measure: Number; unit: Participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 21
Participants
  AEs | 21
  SAEs | 3

2. Secondary Outcome: Mean Number of Seizures
Description: Seizures were episodes of disturbed brain activity that cause changes in attention or behavior. The different types of seizures observed were complex partial, secondarily generalized tonic-clonic, simple partial and others. Mean number of seizures were calculated between each study visit.
Time Frame: Month 6 thereafter every 6 months up to Month 54 or End of Study (EOS) and follow-up (30 days after last dose)
Population: SAS included all participants who had received at least 1 dose of study medication in the open label period. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. Here, 'n' signifies those participants who were evaluable between each visit.
Measure: Mean (Standard Deviation); unit: Seizures
Arm/Group | Pregabalin
Number analyzed (Participants) | 20
Seizures
  Month 6 to Month 12 (n = 20) | 35.10 (46.92)
  Month 12 to Month 18 (n = 18) | 29.70 (26.05)
  Month 18 to Month 24 (n = 19) | 27.80 (28.75)
  Month 24 to Month 30 (n = 18) | 32.50 (33.91)
  Month 30 to Month 36 (n = 18) | 29.30 (29.13)
  Month 36 to Month 42 (n = 17) | 28.70 (28.38)
  Month 42 to Month 48 (n = 11) | 24.80 (32.99)
  Month 54 or EOS (n = 19) | 22.90 (24.57)
  Follow-up (n = 14) | 6.40 (6.39)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Pregabalin
Serious Adverse Events (participants affected / at risk) | 3/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=21)
Lung infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Grand mal convulsion (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=21)
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Cyanosis (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Cerumen impaction (Ear and labyrinth disorders) | 1
Deafness (Ear and labyrinth disorders) | 1
Tympanic membrane perforation (Ear and labyrinth disorders) | 1
Visual acuity reduced (Eye disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Haematochezia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 1
Influenza like illness (General disorders) | 1
Malaise (General disorders) | 1
Ear infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Labyrinthitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 2
Otitis externa (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Back injury (Injury, poisoning and procedural complications) | 1
Epicondylitis (Injury, poisoning and procedural complications) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 10
Foetal exposure during pregnancy (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 2
Hand fracture (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 2
Joint injury (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 4
Limb injury (Injury, poisoning and procedural complications) | 1
Scratch (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Blood iron decreased (Investigations) | 1
Electrocardiogram abnormal (Investigations) | 2
Liver function test abnormal (Investigations) | 1
Vitamin B12 decreased (Investigations) | 1
Vitamin D decreased (Investigations) | 1
Weight decreased (Investigations) | 2
Weight increased (Investigations) | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Balance disorder (Nervous system disorders) | 1
Carotid artery occlusion (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 4
Lethargy (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Anger (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 2
Confusional state (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 1
Mood altered (Psychiatric disorders) | 1
Panic attack (Psychiatric disorders) | 1
Stress (Psychiatric disorders) | 2
Suicidal ideation (Psychiatric disorders) | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
This was a compassionate use study and no formal primary outcome measure was specified a priori. Descriptive safety data were collected, subsequently safety outcome was designated as primary outcome as per National Institute of Health (NIH) criteria.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.